CLINICAL TRIAL: NCT02395380
Title: Evaluation of the Predictive Nature of the Postoperative CRP on Postoperative Recovery in Patients Undergoing Colorectal Resection
Brief Title: Evaluation of the Predictive Nature of the Postoperative CRP on Postoperative Recovery in Patients Undergoing Colorectal Resection (CRP-Track)
Acronym: CRP-Track
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHD 065-14
Record Dates: First submitted 2015-03-02; First posted 2015-03-23 (Estimated); Last update posted 2017-06-19 (Actual); Status verified 2017-06

CONDITIONS: Colorectal Postoperative Complication
Keywords: CRP; Postoperative complication; Length of stay
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- C-reactive protein dosage (Experimental)
  Interventions: Other: C-reactive protein dosage

INTERVENTIONS:
Other: C-reactive protein dosage

SUMMARY:
Colic and rectal resection represents a majority of hospitalizations in visceral surgery. The objective of this study was to evaluate the prognostic of inflammatory markers dosage (CRP, procalcitonin and venous lactate) on the postoperative recovery after colorectal surgery and on the length of stay.

ELIGIBILITY:
Inclusion Criteria:

* Upper age to 18 years
* Planned hospital stay for a colonic resection with anastomosis without permanent or temporary digestive bypass
* Patient with pre-operative CRP lower or egal to 172 mg/L
* No opposition at the participation of the study
* Expected patient return home after surgery (or convalescent home or not medicalized institution)

Exclusion Criteria:

* Patient under guardianship
* Protected or private patient freedom
* Minor patient
* Colectomy surgery with digestive bypass or digestive anastomosis
* Complex combined surgery (significantly intestinal resection associated, another surgical procedure that can interfere with postoperative CRP)
* General inflammatory disease susceptive to modify dosage values
* Anti-inflammatory therapy (AINS/ corticosteroids/ immunosuppressive)
* Patient unable to understand the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2015-07-06 (Actual); Primary Completion 2017-03-11 (Actual); Study Completion 2017-06-13 (Actual)

PRIMARY OUTCOMES:
C-reactive protein rate | 3 postoperative days
  The time of postoperative recovery will be compared to the CRP values at 3 postoperative days.
  The postoperative recovery is a composite endpoint defined by :
  * no pain > 2 on the VAS scale
  * presence of a gaseous bowel
  * patient autonomy in terms of ambulation and body care (IRM 5-6)
  * no fever

CONTACTS AND LOCATIONS:
Overall Officials: Emeric ABET, Study Director — Centre Hospitalier Departemental Vendee
Locations (2):
- France (2):
  - Centre Hospitalier Departemental Vendee, La Roche-sur-Yon
  - CHU Nantes, Nantes